CLINICAL TRIAL: NCT00914719
Title: Alcohol Use and Sexual Risk: An Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution and no subjects enrolled.
Sponsor: University of New Mexico (Other)
Responsible Party: Angela D. Bryan, University of New Mexico
Model: Factorial | Purpose: Prevention
Other Study IDs: R01AA013844-01 (NIH)
Record Dates: First submitted 2009-06-03; First posted 2009-06-05 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Sexual Risk Behavior; Alcohol Use; Drug Use
Keywords: sexual risk behavior among adolescents; alcohol and drug use among adolescents
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol

ARMS (3):
- Information only (Active Comparator)
  Interventions: Behavioral: Information only
- sexual risk reduction intervention (Active Comparator)
  Interventions: Behavioral: Sexual risk reduction intervention
- SRRI+ETOH (Experimental)
  Interventions: Behavioral: sexual risk reduction + alcohol risk reduction component

INTERVENTIONS:
Behavioral: Information only
  Arms: Information only
Behavioral: Sexual risk reduction intervention
  Arms: sexual risk reduction intervention
Behavioral: sexual risk reduction + alcohol risk reduction component
  Arms: SRRI+ETOH

SUMMARY:
Adolescents are at great risk for sexually transmitted diseases (STDs) including the human immunodeficiency virus (HIV) (CDC, 2000a; DiLorenzo & Whaley, 1999). Though the CDC (2000b) reports that overall AIDS incidence is on the decline, there has been no comparable decline in the number of newly diagnosed HIV cases among young people aged 13-19, and young people of color are particularly at risk. Compared to the general adolescent population, adolescents involved with the criminal justice system are younger at first intercourse, have a greater number of sex partners, and lower rates of condom use, resulting in higher rates of unintended pregnancy and STDs (e.g., St. Lawrence et al., 1999). Alcohol use is commonly cited as a reason for lack of condom use among high-risk adolescents such as those involved in the criminal justice system (e.g., Morris et al., 1998) and recent data from our research suggests that it is heavy alcohol use in concert with sexual activity that is most strongly related to lack of condom use (Bryan, Rocheleau, & Robbins, 2002a). The goal of this research is to design, implement, evaluation, and disseminate a successful HIV/STD risk reduction intervention that is theory-based, empirically targeted to adolescents, and articulated to a criminal justice setting. The study compares a sexual risk reduction intervention with a group motivational interviewing alcohol component to a standard sexual risk reduction intervention and a no treatment control condition. The investigators hope to show that: 1) A three-hour one-time intervention has the capacity to reduce sexual risk behavior up to one year post-release among high risk adolescents in detention, 2) A combined sexual and alcohol risk reduction intervention will result in larger decreases in sexual risk behavior than a sexual risk reduction alone, 3) The interventions will exert their effects through changes in mediators derived from a theoretically-based model of condom use intentions and behaviors, and 4) A sexual risk reduction intervention including an alcohol component will be especially effective for those adolescents with higher levels of existing alcohol problems. Finally, given proven efficacy, the intervention curricula and materials will be disseminated for use in adolescent detention facilities throughout the state.

ELIGIBILITY:
Inclusion Criteria:

* All young people between the ages of 14 and 17 who were in the detention centers at which recruitment took place.

Exclusion Criteria:

* Age less than 14 or non-English speaking

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2002-09 (Actual); Primary Completion 2002-09 (Actual); Study Completion 2002-09 (Actual)

PRIMARY OUTCOMES:
Condom use | one year

SECONDARY OUTCOMES:
alcohol use | one year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado, Boulder, Colorado, United States

REFERENCES:
- [Background] Bryan A, Schmiege SJ, Broaddus MR. Mediational analysis in HIV/AIDS research: estimating multivariate path analytic models in a structural equation modeling framework. AIDS Behav. 2007 May;11(3):365-83. doi: 10.1007/s10461-006-9150-2. PMID 16917669
- [Result] Schmiege SJ, Broaddus MR, Levin M, Bryan AD. Randomized trial of group interventions to reduce HIV/STD risk and change theoretical mediators among detained adolescents. J Consult Clin Psychol. 2009 Feb;77(1):38-50. doi: 10.1037/a0014513. PMID 19170452
- [Derived] Bryan AD, Schmiege SJ, Broaddus MR. HIV risk reduction among detained adolescents: a randomized, controlled trial. Pediatrics. 2009 Dec;124(6):e1180-8. doi: 10.1542/peds.2009-0679. Epub 2009 Nov 9. PMID 19901006